CLINICAL TRIAL: NCT01030341
Title: Pilot Study of the Safety, Feasibility, and Potential Efficacy of Continuous Glucose Monitoring and Insulin Pump Therapy in Diabetic Gastroparesis (GLUMIT-DG)
Brief Title: Continuous Glucose Monitoring and Insulin Pump Therapy in Diabetic Gastroparesis
Acronym: GLUMIT-DG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U01DK074008 GLUMIT-DG; U01DK073983 (NIH); U01DK073975 (NIH); U01DK073985 (NIH); U01DK074035 (NIH); U01DK074008 (NIH); U01DK073974 (NIH); U01DK074007 (NIH)
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Gastroparesis
Keywords: Diabetes; Gastroparesis
MeSH Terms: conditions — Diabetes Mellitus; Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CGMS and insulin pump (Experimental): Continuous glucose monitoring in conjunction with insulin pump
  Interventions: Device: CGMS and insulin pump

INTERVENTIONS:
Device: CGMS and insulin pump — Use of continuous glucose monitoring system and insulin pump
  Other Names: Paradigm 722 Insulin pump; Real-Time Continuous Glucose Monitoring System

SUMMARY:
A pilot study to assess the safety, feasibility, and potential (uncontrolled) efficacy of continuous glucose monitoring (CGMS) in conjunction with an insulin pump to improve glycemic control for treatment of type 1 and type 2 diabetic patients with gastroparesis

DETAILED DESCRIPTION:
This multicenter, uncontrolled, open label treatment study is to assess the safety of CGMS in guiding insulin pump therapy for 24 weeks by measuring mild, moderate, and severe hypoglycemic episodes in patients with type 1 and type 2 diabetes and gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years old at registration
* Type 1 or Type 2 diabetes mellitus for at least 2 years
* Symptoms of gastroparesis (nausea, vomiting, early satiety, bloating, fullness, discomfort) for at least 1 year prior to registration
* Gastroparesis Cardinal Symptom Index (GCSI) score of 18
* Delayed gastric emptying on gastric scintigraphy within 1 year of registration, defined as greater than 60% retention at 2 hours or greater than 10% retention at 4 hours
* Hemoglobin A1c of at least 8.0% at registration regardless of current therapy. Individuals already receiving diabetes therapy via an insulin pump will be eligible for study participation if, in the opinion of the investigators, he/she may acquire additional benefit from continuous glucose monitoring that might improve glycemic control
* Normal upper endoscopy within 1 year of registration
* No clinical or imaging evidence of obstruction
* Successful mastering of use of CGMS during the run-in period

Exclusion Criteria:

* Prior gastric surgery including fundoplication
* Other systemic disease potentially causative of gastrointestinal symptoms
* Acute or chronic renal insufficiency with creatinine >1.5 mg/dL
* Psychiatric disease or eating disorder
* Pregnancy
* Any other condition which, in the opinion of the investigators, would impede compliance or hinder completion of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-05; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hamilton, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (7):
- United States (7):
  - California Pacific Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Texas Tech University Health Sciences Center, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/glumit/?query=GLUMIT
URL: https://repository.niddk.nih.gov/studies/glumit/?query=GLUMIT

REFERENCES:
- See also: Click here for information on gastroparesis research — https://jhuccs1.us/gpcrc/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-five patients (age 18-70 years) with diabetes for >2 years in poor glycemic control (HbA1c >8%) with gastroparesis were recruited from 7 centers of the GpCRC from February 2012 through May 2014. Patients had symptoms for >1 year with Gastroparesis Cardinal Symptom Index (GCSI) scores of ≥18.
Pre-assignment Details: Screening Phase-Baseline glycemic profiles were obtained with blinded sensors to acquire >216 hours of glycemic data over 2 weeks.
  Run-In Phase:Participants received detailed instructions in operating the CSII device and had to demonstrate competency in CSII and CGM and electronic CGM data transfer to be enrolled.
Groups:
- All Participants: Continuous glucose monitoring in conjunction with insulin pump
  CGMS and insulin pump: Use of continuous glucose monitoring system and insulin pump
Period: Overall Study
Arm/Group | All Participants
Started | 45 (45 participants met all enrollment criteria by completing the screening and run-in phases)
Completed | 42 (42 participants completed the study)
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 45
Known diabetes duration [Mean (Standard Deviation); unit: years] | 21 (11)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29 (8)
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage] | 9.4 (1.4)
2 hr gastric retention [Mean (Standard Deviation); unit: percentage] | 63 (20)
4 hr gastric retention [Mean (Standard Deviation); unit: percentage] | 32 (20)
GCSI score [Mean (Standard Deviation); unit: units on a scale] — The Gastroparesis Cardinal Symptom Index (GCSI) is the mean of 3 subscales: nausea/vomiting (3 items), post-prandial fullness/early satiety (4 items), and bloating (2 items). Subscale scores were calculated by averaging across items within a subscale. A 6-point Likert scale was used for scoring individual items ranging from 0 (none) to 5 (very severe).
  units on a scale | 3.3 (0.8)
PAGI-QOL [Mean (Standard Deviation); unit: units on a scale] — The Patient Assessment of Upper Gastrointestinal Disorders-Quality of LIfe (PAGI-QOL) contains 30 items with 5 subscales: (1) daily activities; (2) clothing; (3) diet/food habits; (4) relationship; and (5) psychological well-being and distress. Items are scored on a 6-point Likert scale, with response options ranging from 0 (none) to 5 (all of the time). Subscale scores are calculated by averaging the item responses within a each subscale after reversing item scores. A total score is calculated by averaging subscale scores, with higher values indicating improved quality of life.
  units on a scale | 2.4 (1.1)
Volume of Water consumed for water load satiety test [Mean (Standard Deviation); unit: mL] — The Water Load Satiety Test involves drinking cool water over 5 minutes until full. The outcome of interest is the volume of water drank in mL.
  mL | 430 (207)
Volume consumed in a liquid nutrient satiety test [Mean (Standard Deviation); unit: mL] — The liquid nutrient satiety test involves drinking Ensure in 5 minutes until full. The outcome of interest is the amount drank in mL.
  mL | 420 (258)

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemic Episodes
Description: The incidence rate (events / person-week) of mild/moderate (glucose level < 70 mg/dL) and severe (glucose < 50 mg/dL) hypoglycemic episodes during screening vs 24 week of follow-up visits while using a combination of continuous glucose monitoring system (CGMS) and insulin pump therapy.
Time Frame: 4 weeks screening vs 24 weeks follow-up
Population: 44 patients had non-missing data during screening phase and 37 had non-missing data during treatment phase
Measure: Number; unit: event rate per person-week
Arm/Group | All Participants
Number analyzed (Participants) | 44
event rate per person-week
  Screening phase, hypoglycemia / person-week | 1.9
  Treatment phase, hypoglycemia / person-week | 2.2
Statistical Analysis 1: Comparison: All Participants; Null hypothesis: Difference of 0% in the frequencies of hypoglycemic excursions (<50 mg/dL) during the screening phase and treatment phase respectively; Test type: Non-Inferiority or Equivalence — Type I error: 0.05; power: 0.9; p < 0.0001, Regression, Logistic — Threshold for statistical significance: p < 0.05; Generalized estimating equations (GEE) with independent working correlation to account for correlated data comparing screening and treatment phases
Statistical Analysis 2: Comparison: All Participants; Null hypothesis: Difference of 0% in the frequencies of hypoglycemic excursions (<70 mg/dL) during the screening phase and treatment phase respectively; Test type: Non-Inferiority or Equivalence — Type I error: 0.05; power: 0.9; p < 0.0001, Regression, Logistic — Threshold for statistical significance: p < 0.05; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: All Participants; Null hypothesis: Difference of 0% in the frequencies of euglycemic excursions (70-180 mg/dL) during the screening phase and treatment phase respectively; Test type: Non-Inferiority or Equivalence — Type I error: 0.05; power: 0.9; p = 0.005, Regression, Logistic — Threshold for statistical significance: p < 0.05; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: All Participants; Null hypothesis: Difference of 0% in the frequencies of hyperglycemic excursions (>180 mg/dL) during the screening phase and treatment phase respectively; Test type: Non-Inferiority or Equivalence — Type I error: 0.05; power: 0.9; p = 0.04, Regression, Logistic — Threshold for statistical significance: p < 0.05; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: All Participants; Null hypothesis: Difference of 0% in the frequencies of hyperglycemic excursions (>300 mg/dL) during the screening phase and treatment phase respectively; Test type: Non-Inferiority or Equivalence — Type I error: 0.05; power: 0.9; p < 0.0001, Regression, Logistic — Threshold for statistical significance: p < 0.05; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Change in Gastroparesis Cardinal Symptom Index (GCSI) Total and Mean Score and Patient Assessed Gastro-Intestinal Quality of Life (PAGI-QOL) Score
Description: To determine the efficacy of CGMS guided insulin pump therapy on symptoms of gastroparesis as assessed by GCSI total score and mean score and quality of life as assessed by PAGI-QOL score in diabetics with gastroparesis.
  The outcome is assessed using the self-reported total GCSI score, which is computed as the average of the 3 subscores on the GCSI survey: 3-item postprandial fullness/early satiety subscore, the nausea/vomiting subscore (average of 3-items: nausea, retching, vomiting), and bloating subscore (average of 2-items: bloating, stomach visibly larger). Each item is scored from 0 (no) to 5 (very severe) symptoms in the past 2-weeks; the total score ranges from 0 to 5.
  The self-reported PAGI-QOL total score which comprises 30 items scored from 0 (none of the time) to 5 (all of the time) the participant's QOL has been affected in the last 2 weeks.The total score is the mean of the 5 subscale scores and ranges from 0 (lowest QOL) to 5 (highest QOL) in past 2-weeks.
Time Frame: Change from baseline (screening) vs 24 weeks of follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 45
score on a scale
  Change in total GCSI score, screening to 12 weeks | -7.2 (8.2)
  Change in total GCSI score, screening to 24 weeks | -7.1 (9.1)
  Change in GCSI composite, screening to 12 weeks | -0.6 (0.9)
  Change in GCSI composite, screening to 24 weeks | -0.8 (1.0)
  Change in PAGI-QOL score, screening to 12 weeks | 0.7 (0.9)
  Change in PAGI-QOL score, screening to 24 weeks | 0.7 (0.9)
Statistical Analysis 1: Comparison: All Participants; Null hypothesis: No difference in total GCSI score from screening to 12 weeks of treatment; Test type: Non-Inferiority or Equivalence — Mean change = 0; p < 0.0001, paired t-test
Statistical Analysis 2: Comparison: All Participants; Null hypothesis: No difference in total GCSI score from screening to 24 weeks of treatment; Test type: Non-Inferiority or Equivalence — Mean change = 0; p < 0.0001, paired t-test
Statistical Analysis 3: Comparison: All Participants; Null hypothesis: No difference in GCSI composite score from screening to 12 weeks of treatment; Test type: Non-Inferiority or Equivalence — Mean change = 0; p < 0.0001, paired t-test
Statistical Analysis 4: Comparison: All Participants; Null hypothesis: No difference in GCSI composite score from screening to 24 weeks of treatment; Test type: Non-Inferiority or Equivalence — Mean change = 0; p < 0.0001, paired t-test
Statistical Analysis 5: Comparison: All Participants; Null hypothesis: No difference in PAGI-QOL score from screening to 12 weeks of treatment; Test type: Non-Inferiority or Equivalence — Mean change = 0; p < 0.0001, paired t-test
Statistical Analysis 6: Comparison: All Participants; Null hypothesis: No difference in PAGI-QOL score from screening to 24 weeks of treatment; Test type: Non-Inferiority or Equivalence — Mean change = 0; p < 0.0001, paired t-test

ADVERSE EVENTS:
Description: Adverse events were categorized into 3 categories: (1) severe hypoglycemic events, (2) gastroparesis exacerbations which includes nausea, vomiting, abdominal pain and diarrhea and (3) other which includes cholecystectomy, bilateral otitis media, hyperglycemia, rash, dizziness, and retinal detachment.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 16/45
Other Adverse Events (participants affected / at risk) | 12/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | All Participants (N=45)
Severe hypoglycemic events, screening/run-in phase (Metabolism and nutrition disorders) | 2 (2)
Severe hypoglycemic events, treatment phase (Metabolism and nutrition disorders) | 6/42 (6)
Severe hyperglycemic events, treatment phase (Metabolism and nutrition disorders) | 3/42 (3)
Severe gastroparesis exacerbation, screening/run-in phase (Gastrointestinal disorders) | 1 (2)
Severe gastroparesis exacerbation, treatment phase (Gastrointestinal disorders) | 1/42 (1)
Pain, numbness, paresthesia in hands, screening/run-in phase (Nervous system disorders) | 1 (1)
Retinal detachment, screening/run-in phase (Eye disorders) | 1 (1)
Death of unknown cause, screening/run-in phase (General disorders) | 1 (1)
Heart attack, screening/run-in phase (Cardiac disorders) | 1 (1)
Abdominal pain, nausea, vomiting, screening/run-in phase (Gastrointestinal disorders) | 1 (1)
Abdominal pain, nausea, vomiting, treatment phase (Gastrointestinal disorders) | 3/42 (3) — Also included anxiety in one case
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | All Participants (N=45)
Non-severe gastroparesis exacerbation, screening/run-in phase (Gastrointestinal disorders) | 2 (2)
Non-severe gastroparesis exacerbation, treatment phase (Gastrointestinal disorders) | 2/42 (5)
Non-severe hyperglycemia, screening/run-in phase (Metabolism and nutrition disorders) | 1 (1)
Cholecystectomy, screening/run-in phase (Surgical and medical procedures) | 1 (1)
Bilateral otitis externa, treatment phase (Ear and labyrinth disorders) | 1/42 (2) — Also included vomiting and diarrhea in one case
Pruritis/itching rash under CGMS site, screening/run-in phase (Skin and subcutaneous tissue disorders) | 1 (1)
Rash generalized over upper body at CGMS site, treatment phase (Skin and subcutaneous tissue disorders) | 1/42 (1)
Abdominal pain, nausea, vomiting, screening/run-in phase (Gastrointestinal disorders) | 2 (5) — Also included fever, cough, nasal congestion, and/or sore throat in some cases
Abdominal pain, nausea, vomiting, treatment phase (Gastrointestinal disorders) | 2/42 (2) — Also included dizziness, fainting, and/or diarrhea in some cases
Tingling, disorientation, dizziness, screening/run-in phase (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Our sample size and treatment durations were somewhat modest to compare severe hypoglycemic episodes and efficacy outcomes before and during treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No